CLINICAL TRIAL: NCT06554548
Title: A Study Evaluating Food Effect on Pharmacokinetics of HS-10518
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS-10518-103
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Experimental): fasting, fed
  Interventions: Drug: HS-10518
- Sequence BA (Experimental): fed, fasting
  Interventions: Drug: HS-10518

INTERVENTIONS:
Drug: HS-10518 — Treatment A: Single oral dose of HS-10518 160 mg tablet under fasted conditions Treatment B: Single oral dose of HS-10518 160 mg tablet after a high-fat meal

SUMMARY:
The primary objective of this study is to evaluate the effect of food on the pharmacokinetics of HS-10518

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the study procedure，and fully understand the test contents, process and possible adverse reactions, be able to complete the study in accordance with the study regulations.
2. Premenopausal adult female subjects (age ≥18 years old, calculated on the day of signing the informed consent).
3. female subjects weigh at least 45 kg. Body mass index (BMI) = body weight (kg) / height 2 (m2), body mass index is in the range of 18.0 ~ 28.0 (including the critical value).
4. agreed to use effective contraception from signing the informed consent until 3 months after the last dose of medication and not plan to have a child during the study, not plan to donate oocytes within 6 months after the last dose (only nonpharmacologic contraception could be used during the study).

Exclusion Criteria:

1. Her/his Physical examination, vital signs examination, electrocardiogram or clinical laboratory examination, etc., are abnormal and clinically meaningful according to the investigator's judgment.
2. Hepatitis B surface antigen (HBsAg), hepatitis C antibody (anti-HCV), HIV antibody (anti-HCV) HIV antibody (anti-HIV) positive at screening
3. Those with alanine aminotransferase (Alter) and aspartate aminotransferase (Aster) exceeded the upper limit of normal values at screening
4. Those with abnormal and clinically significant ECG results (e.g., QTcF ≥ 450 ms) at screening
5. Those with a prior history of breast cancer, genitourinary cancer, any estrogen-dependent tumor, or any other clinically significant gynecological disease
6. Subjects with a history of osteoporosis
7. Those with a history of migraine, epilepsy, convulsions, depression, or clinically significant depressive state
8. Those with a history of thyroid or parathyroid dysfunction or thyroid-stimulating hormone (TSH), free triiodothyronine (FT3) and free thyroxine (FT4) exceeded the upper limit of normal values at screening
9. Clinically significant gastrointestinal complaints within 7 days before the first dose
10. Those who have a history of severe gastrointestinal diseases (such as Crohn's disease, ulcerative colitis, reflux esophagitis, chronic gastritis, etc.) or a history of surgery that may affect the absorption, distribution, metabolism and excretion of the trial drug (except for simple appendectomy or hernia surgery), and judged by the investigator unsuitable for enrollment
11. Those who have consumed excessive amounts of tea, coffee, and/or caffeinated beverages within 3 months prior to screening (The average is more than 8 cups per day, 1 cup=200 mL)
12. Those who have consumed grapefruit or grapefruit products within 48 hours prior to the first dose.
13. Those who have consumed caffeine-rich and/or xanthine-rich foods or products (such as: coffee, tea, chocolate, and caffeinated carbonated beverages such as cola, etc.), tobacco-containing products (such as cigarettes, etc.), alcohol, or alcoholic products within 48 hours prior to the first dose.
14. Those who drink regularly within 3 months before screening (i.e., drink more than 14 units of alcohol per week, 1 unit = 14 g of alcohol, equivalent to 360 mL of beer or 45 mL of spirits or 150 mL of wine with 40% alcohol, equivalent to drinking 10 bottles of beer or 1 kg of white wine or 3 bottles of red wine per week), or those who cannot stop drinking alcohol products during the study, or those who have a positive alcohol breath test result.
15. Those who smoked more than 5 cigarettes per day on average within 3 months before screening, or those who could not stop using any tobacco products (including e-cigarettes) during the study.
16. Those who have a history of drug abuse, drug dependence, or drug use, or a positive urine screening for drug abuse
17. Those who are prone to allergic reactions, or allergic constitution (such as those who are allergic to pollen, two or more drugs/foods), or those who are known to be allergic to the components of the test drug, and judged by the investigator to be unsuitable for participating in the study.
18. Those who have lost a lot of blood (>400 mL) or donated blood or received blood transfusion within 3 months before screening, or who plan to donate blood during the study period to 1 month after completing the study.
19. Those with a diagnosis of infertility or more than two previous spontaneous abortions.
20. Those with follicle-stimulating hormone (FSH) ≥ 35 U/L at screening.
21. Those who are postpartum, post-abortion or within 6 months after breastfeeding.
22. Those who are pregnant, lactating, or have a positive pregnancy test at screening.
23. Those who have used any drugs (prescription drugs, over-the-counter drugs, Chinese herbal medicines and dietary supplements including vitamins, etc.) within 30 days before the first dose (or at least 7 times the time of the corresponding elimination half-life, whichever is longer)
24. Use of hormonal contraception: those who have used short-acting preparations containing sex hormones (oral, transdermal, intravaginal, etc.) within 3 months before the first dose or long-acting preparations containing sex hormones (any long-acting injections or implants) within 6 months before the first dose.
25. Those who have used the vaccine within 30 days before the first dose or plan to use the vaccine during the study and within 7 days after the end of the study.
26. Those who have participated in other drug clinical trials and used trial drugs within 3 months prior to screening.
27. Those who have unprotected sexual activity within 14 days prior to the first dose.
28. Those who have special dietary requirements and cannot follow a uniform diet.
29. Those who have a history of fainting needle and blood sickness, or who have difficulty in blood collection as assessed by the investigator, or who cannot tolerate venipuncture/indwelling needle blood collection
30. Other circumstances or reasons for which the investigator considered the subject to be unfit to participate in the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Premenopausal adult female subjects
Enrollment: 8 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of HS-10518 | predose and within 48 hours postdose in each treatment period
Area under the plasma concentration versus time curve (AUC0-t) of HS-10518 | within 48 hours postdose in each treatment period
  within 48 hours postdose in each treatment period